CLINICAL TRIAL: NCT05873049
Title: Use of Real-time Fluorescence Imaging in Diabetic Foot Ulcers: A New Strategy to Assess Residual Bacterial Colonization Before Application of Artificial Dermis or Split-thickness Skin Graft
Brief Title: Use of Real-time Fluorescence Imaging in Diabetic Foot Ulcers: the Impact of Colonization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chang shun cheng, Director of Wound Care Center and Department of Plastic Surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N
Record Dates: First submitted 2022-06-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Infection, Surgical Site
Keywords: diabetic foot ulcer; non-infected; autofluorescence; fluorescence imaging; MolecuLight; artificial dermis; split thickness skin graft
MeSH Terms: conditions — Surgical Wound Infection; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fluorescence-guided (Experimental): Patients who used MolecuLight to achieve "high-quality de-colonization" during reconstruction surgery with artificial dermis or split-thickness skin graft
  Interventions: Device: MolecuLight
- Control (No Intervention): Patients who did not use MolecuLight to achieve "high-quality de-colonization" during reconstruction surgery with artificial dermis or split-thickness skin graft

INTERVENTIONS:
Device: MolecuLight — MolecuLight is a handheld fluorescence imaging device that is utilized to help real-time visualize clinically undetectable fluorescent bacteria in wounds. It emits a 405 nm wavelength of safe violet light, which interacts with the wound tissue and bacteria causing certain bacteria to emit red or cyan fluorescence. The fluorescence signals were then captured by MolecuLight and those with bacteria at levels of ≥ 10^4 colony forming units per gram (CFU/g) will be detected and displayed on the screen.
  Arms: Fluorescence-guided

SUMMARY:
The study evaluates the efficacy of fluorescence-guided de-colonization in patients with non-infected diabetic foot ulcers. The efficacy will also be compared between those who used artificial dermis and split-thickness skin graft for reconstruction surgery.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are the main cause of hospitalization in diabetic patients. These hard-to-heal ulcers have a high amputation rate, and a 5-year mortality rate of 50% once being amputated. Treatments for DFU include infection management, wound debridement, revascularization, pressure off-loading, etc. Recently, a novel imaging device called MolecuLight i:X was introduced to help visualize clinically undetectable fluorescent bacteria in wounds and has shown promising effects in the identification of infection. However, as microorganisms almost colonize all chronic wounds, the term "bacterial colonization" should be distinguished from clinical infection. While infection delays the healing process, the impact of colonization on wound reconstruction remains unclear; and the assessment is often more difficult on DFU patients with peripheral neuropathy and vascular diseases. In the present study, investigators will conduct a prospective randomized controlled trial to evaluate the clinical outcome of achieving "high-quality de-colonization" with the aid of MolecuLight i:X in the treatment of noninfected DFU patients, and to compare its efficacy between artificial dermis and split-thickness skin graft.

ELIGIBILITY:
Inclusion Criteria:

1. 20 ≤ age < 80
2. Body mass index (BMI) < 35 kg/m2
3. Glycated hemoglobin (HbA1c) < 10%
4. Target ulcer: (1) 10 ≤ size < 100 cm2 (2)Located on or below malleolus (3)Wagner's grade 2 or 3 initially (4)Margin > 3 cm between target ulcer and other ulcers
5. Transcutaneous oxygen pressure (TcPO2) ≥ 30 mmHg and 0.8 ≤ ankle-brachial index (ABI) ≤ 1.2
6. Patient willingness and signed informed consent

Exclusion Criteria:

1. Pregnancy
2. Type I diabetes mellitus (Type I DM)
3. Active malignancy
4. Taking glucocorticoids, immunosuppressants, or in an immunocompromised status
5. Lab test upon admission for reconstruction surgery: (1) hemoglobin (Hb) < 8.0 g/dL, or white blood cell (WBC) < 3000 cell/μg (2) aspartate aminotransferase (AST) / alanine aminotransferase (ALT) / total bilirubin > 3x upper normal limits (3) albumin < 2.5 g/dL

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete healing time | 180 days after reconstruction surgery
  The time for complete wound epithelialization or closure without drainage after reconstruction surgery.
Wound healing rate on 30, 60, 90 and 180 days | 180 days after reconstruction surgery
  The healing percentage of wound 30, 60, 90 and 180 days after reconstruction surgery.
Artificial dermis (AD) or split-thickness skin graft (STSG) take rate | 21 days after reconstruction surgery
  The take percentage of artificial dermis or split-thickness skin graft 21 days after reconstruction surgery.

SECONDARY OUTCOMES:
Percentage of bacteria before MolecuLight de-colonization | Immediately after last debridement
  The percentage of bacteria after the last debridement without using MolecuLight to do de-colonization.
Percentage of bacteria after MolecuLight de-colonization | Immediately after de-colonization with MolecuLight
  The percentage of bacteria after using MolecuLight to do de-colonization.
Wound surface area on 30, 60, 90 and 180 days | 30, 60, 90 and 180 days after reconstruction surgery
  The surface area of wound 30, 60, 90 and 180 days after reconstruction surgery.
Reasons for poor AD or STSG take rate | 21 days after reconstruction surgery
  Reasons for poor take rate of artificial dermis or split-thickness skin graft 21 days after reconstruction surgery may include as follows: (1) weak graft fixation (2) seroma (3) hematoma (4) wound localized infection (5) osteomyelitis (6) irreversible ischemic ulcers (7) systemic cause
Complications on 180 days | 180 days after reconstruction surgery
  Complications evaluated 180 days after reconstruction surgery may include as follows: (1) wound recurrence (2) higher-level amputation (3) above or below knee amputation (4) vascular restenosis (5) mortality
Vancouver scar score on 180 days | 180 days after reconstruction surgery.
  The vancouver scar score of wound evaluated 180 days after reconstruction surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Shun-Cheng Chang, Director, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital First Medical Building, New Taipei City, Taiwan